CLINICAL TRIAL: NCT02696096
Title: Neuroimaging Predictors of Relapse During Treatment for Opiate Dependence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Butler Hospital (Other)
Responsible Party: Principal Investigator, Michael Stein, MD, Principle Investigator, Butler Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 793387
Record Dates: First submitted 2016-02-09; First posted 2016-03-02 (Estimated); Results first posted 2022-08-17 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-07

CONDITIONS: Opioid Addiction
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination; Buprenorphine

ARMS (1):
- All Participants (Other): FMRI Suboxone
  Interventions: Other: FMRI; Drug: Suboxone

INTERVENTIONS:
Other: FMRI — all participants will complete 2 FMRIs
  Other Names: functional magnetic resonance imaging
Drug: Suboxone — all participants will be prescribed Suboxone for 4 months during their study participation
  Other Names: buprenorphine

SUMMARY:
This study proposes to use functional magnetic resonance imaging (FMRI) to observe brain activity and behavior associated with decision-making about rewards (DD task), working memory and working memory cognitive persistence (WM task), and craving (CR task) in 72 opiate dependent participants initiating buprenorphine. While stably using opiates (initial study appointment) and again during withdrawal (approximately 3 days later), participants will receive an FMRI scan with behavioral challenges; immediately after the second FMRI, they will receive their first dose of buprenorphine. Buprenorphine treatment will continue for twelve weeks, followed by a four week taper. Urine toxicological analysis will be performed prior to the first scanning session, weekly for two weeks and biweekly thereafter.

Participation for all individuals will last 4 months. Assessments will occur at baseline, and weeks 1, 2, 4, 8, and 12. Buprenorphine induction will begin at the completion of the second scan; follow-up medical visits will align with study assessments on weeks 1, 2, 4, 8 and 12. All participants will receive 16 weeks of buprenorphine (the final 4 of these 16 weeks will include a taper).

ELIGIBILITY:
Inclusion Criteria:

* opiate dependent persons
* 21-50 years old
* interested in initiating outpatient buprenorphine treatment

Exclusion Criteria:

* current methadone maintenance treatment program participation
* medically necessary prescription opiate treatment (e.g., for chronic pain)
* current criteria for a DSM-V diagnosis of substance dependence for sedative or hypnotic drugs, alcohol, stimulants, cocaine, inhalants, hallucinogens
* diagnosis of organic brain disorder, bipolar disorder, schizophrenia, schizo-affective, schizophreniform or paranoid disorder
* current suicidality on the Modified Scale for Suicidal Ideation
* evidence of neuropsychological dysfunction as assessed by the study physician with confirmation with the Folstein Mini-Mental Status Examination•
* anticipated major painful event (significant surgical procedure) in the coming 4 months
* probation or parole requirements or an upcoming move that might interfere with protocol participation
* history of allergic reaction to buprenorphine or naloxone
* currently pregnant or planning to become pregnant in the next 4 months
* history of neurological disorder (e.g., epilepsy, stroke, brain injury)
* impaired uncorrected vision
* FMRI contraindications (e.g., claustrophobia, specific metallic implants and injuries)

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants Who Used Illicit Opioids and Were Interested in Transitioning to Buprenorphine: All participants completed 2 fMRI's and induction on Buprenorphine during the baseline enrollment. Participants were provided Buprenorphine and completed assessments for 4 months. Opioid abstinence was monitored through self-report and urine toxicology during the study period.
Period: Overall Study
Arm/Group | Participants Who Used Illicit Opioids and Were Interested in Transitioning to Buprenorphine
Started | 21
Opioid Abstinence During Study Period | 11
Completed | 19
Not Completed | 2
Not completed — ruled out at screening | 1
Not completed — did not attend second fMRI | 1

BASELINE CHARACTERISTICS:
Population: Participants were using illicit opioids and seeking Buprenorphine treatment.
Arm/Group | All Participants
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.63 (7.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 14
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Changes in Resting State Disorganization Between Baseline and One Week by Person by Lapsed Category
Description: The measure of resting state organization is a z-value derived from Pearson's r-values. They represent the effect of the association between the brain activity of the seed region and each brain voxel over time during the resting state FMRI scan. A central z-value of 0 means that there is no association between the seed region and the voxel.
  Positive and negative z-values approaching 0 reflect increasingly weaker associations, and more extreme positive and negative values reflect stronger associations. Attributing the qualitative labels better or worse to these values depend upon the brain network and context. In many networks (eg, task-positive cognitive control network), a stronger positive correlation is thought to reflect better network organization. In the task-negative default mode network a stronger positive relationship is considered by some as worse. For this study, these are not yet used as clinical measures and there are not known cutoffs.
Time Frame: Baseline and 1 week
Population: Mean fMRI resting state disorganization at baseline among no-lapse and lapse groups
Measure: Mean (Standard Deviation); unit: Mean default mode network (DMN) z-scores
Groups:
- No Lapse: No opioid use during the study period
- Lapse: Opioid use during the study period
Arm/Group | No Lapse | Lapse
Number analyzed (Participants) | 6 | 5
Mean default mode network (DMN) z-scores
  DMN synchrony active use | 0.315 (0.057) | 0.328 (0.076)
  DMN synchrony abstinent | 0.384 (0.098) | 0.394 (0.139)

2. Primary Outcome: Working Memory - Between Groups at Baseline by Lapsed Category
Description: fMRI working memory differences between participants who lapse back to opioid use and those who don't
Time Frame: Baseline
Population: Mean fMRI working memory response at baseline among no-lapse and lapse groups
Measure: Mean (Standard Deviation); unit: % fMRI signal change
Arm/Group | No Lapse | Lapse
Number analyzed (Participants) | 9 | 7
% fMRI signal change
  bilateral SMA | 0.45 (0.14) | 0.42 (0.27)
  R middle frontal gyrus | 0.39 (0.15) | 0.40 (0.23)
  R inferior parietal lobule | 0.34 (0.14) | 0.33 (0.24)
  L inferior parietal lobule | 0.36 (0.14) | 0.32 (0.25)
  L middle frontal gyrus (a) | 0.46 (0.20) | 0.49 (0.26)
  L middle frontal gyrus (b) | 0.36 (0.16) | 0.33 (0.25)
  L middle frontal gyrus (c) | 0.39 (0.22) | 0.36 (0.28)
  bilateral precuneus | 0.38 (0.20) | 0.37 (0.26)
  R anterior insula | 0.42 (0.14) | 0.39 (0.26)

3. Primary Outcome: Changes in Working Memory - Within Groups During Satiation and Withdrawal
Description: fMRI working memory differences under satiation vs withdrawal from opioids
Time Frame: Baseline and 1 week
Population: Within-group analyses contrasting two fMRI responses
Measure: Mean (Standard Deviation); unit: % fMRI signal change
Groups:
- fMRI During Withdrawal: this fMRI was completed when the participants were experiencing opioid withdrawal symptoms
- fMRI During Opioid Use: this fMRI was completed while participants were satiated with opioids
Arm/Group | fMRI During Withdrawal | fMRI During Opioid Use
Number analyzed (Participants) | 12 | 12
% fMRI signal change
  Mean Brain Response in R middle frontal gyrus | 0.35 (0.30) | 0.37 (0.25)
  Mean Brain Response in R inferior parietal lobule | 0.33 (0.29) | 0.42 (0.22)
  Mean Brain Response in L inferior parietal lobule | 0.47 (0.43) | 0.54 (0.32)
  Mean Brain Response in bilateral supplementary motor | 0.34 (0.27) | 0.35 (0.22)

ADVERSE EVENTS:
Time Frame: 4 months
Description: Adverse events were as noted in clinicaltrials.gov
Arm/Group | No Lapse | Lapse
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/7
Other Adverse Events (participants affected / at risk) | 0/12 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-06-22): https://cdn.clinicaltrials.gov/large-docs/96/NCT02696096/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-22): https://cdn.clinicaltrials.gov/large-docs/96/NCT02696096/SAP_001.pdf